CLINICAL TRIAL: NCT02475941
Title: Early Weight Bearing on Supracondylar Distal Femur Fractures in Elderly Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Louis University (Other)
Responsible Party: Principal Investigator, Howard Place, MD, Professor, Department of Orthopaedic Surgery, St. Louis University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24664
Record Dates: First submitted 2015-06-04; First posted 2015-06-19 (Estimated); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Distal Femur Fractures
Keywords: geriatric fractures
MeSH Terms: conditions — Femoral Fractures, Distal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early Weight Bearing (Experimental): Surgeon based prospective cohort supported in the literature to answer research questions in which surgeons have a preferred treatment type. Early weight bearing are those who are permitted in the post operative instructions to be Weight Bear as tolerated after fracture fixation.
  Interventions: Other: Early Weight Bearing
- Non Weight Bearing (Active Comparator): Surgeon based prospective cohort supported in the literature to answer research questions in which surgeons have a preferred treatment type. Non weight bearing are those who are NOT permitted in the post operative instructions to be Weight Bear after fracture fixation.
  Interventions: Other: Non Weight bearing

INTERVENTIONS:
Other: Non Weight bearing — The design will be a surgeon based prospective cohort supported in the literature to answer research questions in which surgeons may have a preferred treatment type. Each surgeon will treat study subjects by his or her single chosen method (weight bearing as tolerated post operatively versus non weight bearing).
  The benefits of early weight bearing are accelerated functional recovery, increased independence, decreased impact on the family, increased psychological benefits, reduced use of healthcare resources, decreased need for family intervention, and family to take care of the patient.
  Arms: Non Weight Bearing
Other: Early Weight Bearing — The design will be a surgeon based prospective cohort supported in the literature to answer research questions in which surgeons may have a preferred treatment type. Each surgeon will treat study subjects by his or her single chosen method (weight bearing as tolerated post operatively versus non weight bearing).
  The benefits of early weight bearing are accelerated functional recovery, increased independence, decreased impact on the family, increased psychological benefits, reduced use of healthcare resources, decreased need for family intervention, and family to take care of the patient.
  Arms: Early Weight Bearing

SUMMARY:
The investigators will be looking at geriatric distal femur fractures. The investigators will prospectively enroll these patients and allow patients to either weight bear as tolerated or limit their weight bearing post operatively. The investigators will evaluate functional outcomes.

DETAILED DESCRIPTION:
Supracondylar femur fractures represent 4-7% of femur fractures. These are a common orthopaedic injury with an overall incidence of 37 per 100,000 person-years. These fractures are complex and challenging for orthopaedic surgeons. The fracture needs to be correctly reduced and, like nearly all fractures, fixed with enough stability to permit early joint motion. This allows for earlier patient rehabilitation, which can improve outcomes. There are a number of different fixation devices. Fixed angle implants such as retrograde intramedullary nails, angled blade plates, and 95-degree side plates have had good clinical outcomes with resistance to varus collapse. Recently, locking plates have become the standard method for distal femoral fracture fixation. Hendersen et al. provided a systematic review of locking plate fixation and demonstrated the range of complications as 0% to 32% and implant failure occurring late with 75% of failures occurring after 3 months and 50% occurring after 6 months. Ricci et al. sought to determine risk factors associated with failure of locked plate fixation of distal femur fractures and found that 19% required reoperation. The risk factors for reoperation found in this study were diabetes, smoking, increased body mass index, shorter plate length and open fracture. Most factors are out of surgeon control but are important to evaluate when considering prognosis.

After the fracture has been open reduced and internally fixed, there is debate on postoperative management of weight bearing. Weight bearing following fixation is generally restricted for 6 to 12 weeks until radiologic evidence of evidence demonstrates sufficient callous. This restricted weight bearing is primarily due to concerns of implant failure and loss of reduction. A study by Brumback et al. examined intramedullary nail fixation of distal femur fractures and concluded to allow full weight bearing of comminuted femoral shaft fractures with antegrade intramedullary nail. This study led surgeons to accelerate their rehabilitation protocols.

The post-operative weight bearing recommendations for distal femur fractures treated with locking plate vary widely which motivated Granata et al. to evaluate the biomechanics of immediate weight bearing of distal femur fractures treated with locked plate fixation. They found that the fatigue limit of the locked plate constructs was 1.9 times body weight for an average 70-kilogram patient over a simulated 10-week postoperative course. Although this study could not fully support immediate weight bearing due to the fact that femoral loads during gait have been estimated to be around 2 times body weight, it demonstrated adequate hardware fixation with weight bearing.

The benefits of early weight bearing are accelerated functional recovery, increased independence, decreased impact on the family, increased psychological benefits, reduced use of healthcare resources, decreased need for family intervention, and family to take care of the patient. The downside is the strength of fixation, the risk of implant failure, and the risk of loss of reduction. The goals are to evaluate the fracture, the complication rate, the mortality rate, and the risks of healthcare resources that have been used.

ELIGIBILITY:
Inclusion Criteria:

* Distal femur fractures, including periprosthetic fractures
* AO/OTA classification 33
* Above 64 years of age and below 90 years of age
* Household ambulators: defined as an individual who can walk continuously for distances that are considered reasonable for walking inside the home but limited for walking in the community due of endurance, strength, or safety concerns

Exclusion Criteria:

* Those who do not fit the inclusion criteria
* Concomitant ipsilateral lower extremity injury
* Contralateral lower extremity injury.
* Vascular injury of concomitant lower extremity requiring repair
* Pathologic fracture
* Definitive treatment delay of more than 2 weeks from initial injury
* Unable to comply with post-operative rehabilitation protocols or instructions
* Current or impending incarceration

Ages: 64 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-05-11 (Actual); Primary Completion 2019-01-02 (Actual); Study Completion 2019-09-27 (Actual)

PRIMARY OUTCOMES:
Fracture Healing in Early Weight Bearing assessed by radiographs | Post op-3 months
  Will assess radiographs to assess for a healed fracture with no loss of fixation or need for secondary surgery

SECONDARY OUTCOMES:
Visual Analog Scale to assess pain | Pre-injury function and at 6 weeks, 3, 6 and 12 months post-injury
  Assess pain to compare between two groups
Oxford Knee Score to measure knee function | Pre-injury function and at 6 weeks, 3, 6 and 12 months post-injury
  Validated outcome measure to document knee function to compare between two groups
SF12 to measure return to function | Pre-injury function and at 6 weeks, 3, 6 and 12 months post-injury
  Measures patients outcome based on their return to function.

CONTACTS AND LOCATIONS:
Overall Officials: Howard Place, MD, Principal Investigator — St. Louis University
Locations (6):
- United States (6):
  - Wellstar, Atlanta, Georgia
  - St. Louis Medical Center, St Louis, Missouri
  - Duke University, Durham, North Carolina
  - Wake Forest University, Winston-Salem, North Carolina
  - Grennville Health Sysytems, Greenville, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee

REFERENCES:
- [Result] Nieves JW, Bilezikian JP, Lane JM, Einhorn TA, Wang Y, Steinbuch M, Cosman F. Fragility fractures of the hip and femur: incidence and patient characteristics. Osteoporos Int. 2010 Mar;21(3):399-408. doi: 10.1007/s00198-009-0962-6. Epub 2009 May 30. PMID 19484169
- [Result] Zlowodzki M, Bhandari M, Marek DJ, Cole PA, Kregor PJ. Operative treatment of acute distal femur fractures: systematic review of 2 comparative studies and 45 case series (1989 to 2005). J Orthop Trauma. 2006 May;20(5):366-71. doi: 10.1097/00005131-200605000-00013. PMID 16766943
- [Result] David SM, Harrow ME, Peindl RD, Frick SL, Kellam JF. Comparative biomechanical analysis of supracondylar femur fracture fixation: locked intramedullary nail versus 95-degree angled plate. J Orthop Trauma. 1997 Jul;11(5):344-50. doi: 10.1097/00005131-199707000-00008. PMID 9294798
- [Result] Christodoulou A, Terzidis I, Ploumis A, Metsovitis S, Koukoulidis A, Toptsis C. Supracondylar femoral fractures in elderly patients treated with the dynamic condylar screw and the retrograde intramedullary nail: a comparative study of the two methods. Arch Orthop Trauma Surg. 2005 Mar;125(2):73-9. doi: 10.1007/s00402-004-0771-5. Epub 2004 Dec 21. PMID 15611863
- [Result] Hartin NL, Harris I, Hazratwala K. Retrograde nailing versus fixed-angle blade plating for supracondylar femoral fractures: a randomized controlled trial. ANZ J Surg. 2006 May;76(5):290-4. doi: 10.1111/j.1445-2197.2006.03714.x. PMID 16768683
- [Result] Ricci WM, Streubel PN, Morshed S, Collinge CA, Nork SE, Gardner MJ. Risk factors for failure of locked plate fixation of distal femur fractures: an analysis of 335 cases. J Orthop Trauma. 2014 Feb;28(2):83-9. doi: 10.1097/BOT.0b013e31829e6dd0. PMID 23760176
- [Result] Henderson CE, Kuhl LL, Fitzpatrick DC, Marsh JL. Locking plates for distal femur fractures: is there a problem with fracture healing? J Orthop Trauma. 2011 Feb;25 Suppl 1:S8-14. doi: 10.1097/BOT.0b013e3182070127. PMID 21248560
- [Result] Forster MC, Komarsamy B, Davison JN. Distal femoral fractures: a review of fixation methods. Injury. 2006 Feb;37(2):97-108. doi: 10.1016/j.injury.2005.02.015. Epub 2005 Apr 25. PMID 16439229
- [Result] Kregor PJ, Stannard JA, Zlowodzki M, Cole PA. Treatment of distal femur fractures using the less invasive stabilization system: surgical experience and early clinical results in 103 fractures. J Orthop Trauma. 2004 Sep;18(8):509-20. doi: 10.1097/00005131-200409000-00006. PMID 15475846
- [Result] Markmiller M, Konrad G, Sudkamp N. Femur-LISS and distal femoral nail for fixation of distal femoral fractures: are there differences in outcome and complications? Clin Orthop Relat Res. 2004 Sep;(426):252-7. doi: 10.1097/01.blo.0000141935.86481.ba. PMID 15346082
- [Result] Brumback RJ, Toal TR Jr, Murphy-Zane MS, Novak VP, Belkoff SM. Immediate weight-bearing after treatment of a comminuted fracture of the femoral shaft with a statically locked intramedullary nail. J Bone Joint Surg Am. 1999 Nov;81(11):1538-44. doi: 10.2106/00004623-199911000-00005. PMID 10565645
- [Result] Granata JD, Litsky AS, Lustenberger DP, Probe RA, Ellis TJ. Immediate weight bearing of comminuted supracondylar femur fractures using locked plate fixation. Orthopedics. 2012 Aug 1;35(8):e1210-3. doi: 10.3928/01477447-20120725-21. PMID 22868607
- [Result] McGraw P, Kumar A. Periprosthetic fractures of the femur after total knee arthroplasty. J Orthop Traumatol. 2010 Sep;11(3):135-41. doi: 10.1007/s10195-010-0099-6. Epub 2010 Jul 27. PMID 20661762
- [Result] Weinstein AM, Rome BN, Reichmann WM, Collins JE, Burbine SA, Thornhill TS, Wright J, Katz JN, Losina E. Estimating the burden of total knee replacement in the United States. J Bone Joint Surg Am. 2013 Mar 6;95(5):385-92. doi: 10.2106/JBJS.L.00206. PMID 23344005